CLINICAL TRIAL: NCT04856059
Title: Fabry Cardiomyopathy: Identification of Early Myocardial Structural and Tissue Abnormalities Using Multiparametric MRI
Acronym: FIESTA-MRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Vancouver General Hospital (Other); The Cleveland Clinic (Other); Icahn School of Medicine at Mount Sinai (Other); Mayo Clinic (Other); University of Colorado, Denver (Other); IRCCS Policlinico S. Donato (Other); Alberta Health services (Other); Libin Cardiovascular Institute of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-5167
Record Dates: First submitted 2021-04-20; First posted 2021-04-22 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Fabry Disease
Keywords: Fabry disease; Fabry cardiomyopathy; cardiac MRI; CMR; T1 mapping; T2mapping
MeSH Terms: conditions — Fabry Disease | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Intervention Model Description: cardiac MRI
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac MRI, ECG and Blood Biomarkers (Other): Additional sequences will be performed during routine clinical cardiac MRI and additional blood samples will be collected during routine blood work.
  Interventions: Diagnostic Test: Cardiac MRI, ECG/Holter and Blood Biomarkers

INTERVENTIONS:
Diagnostic Test: Cardiac MRI, ECG/Holter and Blood Biomarkers — Cardiac MRI including T1/T2 mapping, ECG and blood biomarker evaluation will be performed at baseline and follow-up

SUMMARY:
This study will evaluate whether cardiac MRI T1 and T2 mapping improves our ability to detect early abnormalities in the heart in patients with Fabry disease and identify patients at increase risk of adverse events.

DETAILED DESCRIPTION:
Fabry disease is an inherited disorder that affects many organs in the body, including the heart. Men and women are both affected, with average life expectancy reduced by 10-20 years. The heart muscle can become thick and scarred in over half of patients, eventually resulting in heart failure, abnormal rhythm and death. The focus of this study will be on improving the detection of early heart disease before irreversible damage has occurred in order to improve patient outcomes.

It is hypothesized that new cardiac MRI techniques called T1 and T2 mapping will improve the ability to detect early abnormalities in the heart. Early detection of cardiac disease may enable a personalized treatment approach, potentially improving patient outcomes. The results of the study will identify which patients might benefit from early initiation of treatment to prevent bad outcomes in the future by using cardiac MRI to identify those at higher risk.

ELIGIBILITY:
Inclusion Criteria:

* Fabry disease;
* Age ≥ 18 years.

Exclusion Criteria:

* History of myocardial infarction;
* Contraindication to MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | 5 years
  MACE will be assessed as a composite endpoint defined by the development on one or more of events such as sustained ventricular tachycardia (VT), severe bradycardia, heart failure hospitalization and cardiac death.

SECONDARY OUTCOMES:
The FAbry STabilization indEX (FASTEX) score | 3 years
  FAbry STabilization indEX (FASTEX) score will be evaluated to assess clinical stability or progression of Fabry disease at follow-up.
  FASTEX score change of ≥20% will be considered an indication of clinical worsening at follow-up.
  Minimum value 0%. No maximum value. Higher score change indicates worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Hanneman, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No